CLINICAL TRIAL: NCT07292987
Title: Implementation and Evaluation of a Post-diagnostic Announcement Protocol at the CRMR RefeRet of the Quinze-Vingts National Ophthalmology Hospital
Brief Title: Implementation and Evaluation of a Post-Diagnostic Announcement Protocol at the CRMR RefeRet, Quinze-Vingts Hospital
Acronym: RP-DIAG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: P25-02; 2025-A01308-41 (Other: ANSM)
Record Dates: First submitted 2025-11-25; First posted 2025-12-18 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Retinitis Pigmentosa (RP)
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual care group (Active Comparator)
  Interventions: Behavioral: Usual Care
- Enhanced care group (Experimental)
  Interventions: Behavioral: Enhanced post-diagnostic support

INTERVENTIONS:
Behavioral: Enhanced post-diagnostic support — Nurse-led and psychologist consultation
  Arms: Enhanced care group
Behavioral: Usual Care — Standard ophthalmologist consultation with optional psychologist consultation
  Arms: Usual care group

SUMMARY:
This study explores whether adding early nurse-led and psychological support after the diagnosis of retinitis pigmentosa (RP) can improve patient experience and emotional well-being. RP is a rare, progressive eye disease often diagnosed after a long and difficult process, and receiving the diagnosis can be emotionally distressing.

Eighty newly diagnosed adults will be randomly assigned to either usual care or an enhanced pathway that includes early follow-up with a nurse, structured emotional monitoring, and a psychologist visit at six months.

The study aims to determine if this structured support improves patient satisfaction and reduces anxiety and depression compared with standard care.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is a rare genetic disease causing progressive vision loss. The announcement of diagnosis is a key moment that may trigger anxiety or depression, yet post-diagnostic care in ophthalmology often remains limited to medical information.

This prospective, monocentric, randomized study at the Quinze-Vingts National Ophthalmology Hospital tests a structured post-diagnostic support pathway that combines early nurse-led follow-up and systematic psychological support.

Eighty newly diagnosed patients aged 18-65 will be randomized into two parallel groups. The experimental group will receive early nurse consultations at 15 days and 6 months, psychological follow-up at 6 months, and repeated HADS assessments. The control group will receive usual care.

The primary outcome is patient satisfaction at 12 months (PREM). Secondary outcomes include changes in anxiety and depression (HADS) and feasibility feedback from nursing staff (RETEX).

Findings will inform the design of sustainable, multidisciplinary care models for rare eye diseases.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with retinitis pigmentosa (RP) and followed at the Quinze-Vingts Rare Eye Disease Center, with diagnosis made after the project begins
* Aged 18 to 65 years
* Male or female
* French-speaking
* Have a phone number
* Reside in France

Exclusion Criteria:

* Pregnant women
* Participants enrolled in a therapeutic clinical trial within the past 12 months
* Individuals deprived of liberty by judicial or administrative decision
* Adults under legal protection or unable to provide informed consent
* Individuals with other medical conditions or taking treatments that could interfere with study evaluations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction via PREM at 12 months | 12 months
  Difference in patient satisfaction via PREM (Patient Reported Experience Measure) at 12 months between the two arms. Items were rated on a 5-point Likert scale ranging from 1 (extremely worse than expected) to 5 (better than expected). Higher scores indicate a better perceived quality of care and psychological support.

SECONDARY OUTCOMES:
Psychological impact after post-diagnostic support via HADS | 15 days, 6 months and 12 months after diagnosis
  Evaluation of the psychological impact of the enhanced post-diagnostic care. Longitudinal assessment of emotional well-being in the experimental group will be performed using the Hospital Anxiety and Depression Scale (HADS) at three key time points. Each subscale (anxiety and depression) ranges from 0 to 21, with higher scores indicating greater symptom severity (worse outcome).
Feasibility and staff experience of implementing enhanced post-diagnostic support via RETEX and observation log | 15 days, 6 months and 12 months after diagnosis
  Nursing staff will complete a RETEX (Retour d'Expérience) questionnaire to assess the feasibility of the enhanced post-diagnostic care. The questionnaire evaluates challenges such as physician presence, adequacy of tools and setting, respect for patient privacy, communication with other staff, and consultation duration. The RETEX questionnaire consists of 11 dichotomous (Yes/No) items completed by nursing staff. Total score ranges from 0 to 11. Higher scores indicate greater perceived emotional and/or organizational burden, whereas lower scores indicate better feasibility and professional comfort.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Audo, Pr, Principal Investigator — CRMR Centre Hospitalier National D' Ophtalmologie Des Quinze-Vingts
Locations (1):
- Centre Hospitalier National D' Ophtalmologie Des Quinze-Vingts, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT07292987/Prot_000.pdf